CLINICAL TRIAL: NCT00058123
Title: A Phase II Trial of Poly ICLC in Patients With Recurrent Anaplastic Glioma
Brief Title: Poly-ICLC in Treating Patients With Recurrent or Progressive Anaplastic Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABTC-0106 CDR0000287012; U01CA062399 (NIH); NABTC-0106
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult mixed glioma; adult anaplastic oligodendroglioma; recurrent adult brain tumor; adult anaplastic ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioma; Oligodendroglioma; Brain Neoplasms; Ependymoma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Poly-ICLC Recurrent gliomas (Experimental): Poly-ICLC 20ug/kg 3 times a week 4 week cycles (Monday-Wednesday-Friday)
  Intramuscular injection
  Drug Poly-ICLC
  Interventions: Drug: poly ICLC

INTERVENTIONS:
Drug: poly ICLC

SUMMARY:
RATIONALE: Biological therapies such as poly-ICLC use different ways to stimulate the immune system and stop tumor cells from growing.

PURPOSE: This phase II trial is studying how poly-ICLC works in treating patients with recurrent, progressive, or relapsed anaplastic glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with recurrent or progressive anaplastic glioma treated with poly ICLC.
* Determine the efficacy of this drug, in terms of 6-month progression-free survival, in these patients.
* Determine the safety profile of this drug in these patients.
* Determine the survival of patients treated with this drug.
* Determine the tumor response rate in patients treated with this drug.
* Determine the biological effects of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive poly ICLC intramuscularly 3 times a week for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 22-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial anaplastic glioma, including any of the following subtypes:

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Other anaplastic gliomas NOTE: Patients with an original histology of low-grade glioma are allowed provided a subsequent histological diagnosis of an anaplastic glioma is made
* Must have evidence of tumor recurrence or progression by MRI or CT scan* NOTE: *Steroid dose must be stable for at least 5 days before scan
* Prior radiotherapy required

  * Patients who have had prior interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis by positron-emission tomography, thallium scanning, magnetic resonance spectroscopy, or surgical documentation of disease
* Relapsed disease

  * Progression after initial therapy (e.g., radiotherapy with or without chemotherapy)
  * No more than 3 prior therapies (initial therapy and treatment for no more than 2 prior relapses)
  * Surgical resection for relapsed disease with no anticancer therapy for up to 12 weeks followed by another surgical resection is considered 1 relapse
  * For patients who have had prior therapy for a low-grade glioma, the surgical diagnosis of high-grade glioma is considered the first relapse
* Must be registered in the North American Brain Tumor Consortium Data Management Center database

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic

* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN

Renal

* Creatinine less than 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other cancer within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection
* No concurrent serious medical illness
* No significant medical illness that cannot be adequately controlled with therapy or that would preclude tolerability of study drug
* No disease that would obscure toxicity or dangerously alter drug metabolism

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 1 week since prior interferon or thalidomide
* No prior poly ICLC

Chemotherapy

* See Disease Characteristics
* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 1 week since prior tamoxifen

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* Recovered from all prior therapy
* At least 1 week since other prior noncytotoxic agents (e.g., isotretinoin), excluding radiosensitizers
* At least 4 weeks since prior cytotoxic therapy
* At least 4 weeks since prior investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-03-07 (Actual); Primary Completion 2007-10-06 (Actual); Study Completion 2009-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Chang, MD, Study Chair — University of California, San Francisco
Locations (8):
- United States (8):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Butowski N, Lamborn KR, Lee BL, Prados MD, Cloughesy T, DeAngelis LM, Abrey L, Fink K, Lieberman F, Mehta M, Ian Robins H, Junck L, Salazar AM, Chang SM. A North American brain tumor consortium phase II study of poly-ICLC for adult patients with recurrent anaplastic gliomas. J Neurooncol. 2009 Jan;91(2):183-9. doi: 10.1007/s11060-008-9705-3. Epub 2008 Oct 11. PMID 18850068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 patients enrolled between 7/14/2003 and 12/192005 at Outpatient Clinical Centers
Groups:
- Poly-ICLC Recurrent Gliomas: Poly-ICLC 20ug/kg 3 times a week 4 week cycles (Monday-Wednesday-Friday)
  Intramuscular injection
  poly ICLC
Period: Overall Study
Arm/Group | Poly-ICLC Recurrent Gliomas
Started | 55
Completed | 45
Not Completed | 10
Not completed — Wrong histology | 9
Not completed — Received >3 prior treatments | 1

BASELINE CHARACTERISTICS:
Population: 55 enrolled however, 10 were not evaluable for outcomes
Arm/Group | Poly-ICLC Recurrent Gliomas
Number analyzed (Participants) | 45
Age, Customized [Median (Full Range); unit: years] | 43 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
Karnofsky Performance Status Scale [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 90 [60 to 100]
Histology [Number; unit: participants] — WHO Classification
  participants
    Anaplastic Astrocytoma | 32
    Anaplastic Oligodendroglioma | 10
    Anaplastic Mixed Oligoastrocytoma | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Objective Response Rate (ORR)
Description: Measurable: Bidimensionally measurable lesions w/ clearly defined margins by MRI Evaluable: Unidimensionally measurable lesions, masses w/margins not clearly defined.
  Complete Response (CR): Complete disappearance of all measurable/evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients on minimal/no steroids.
  Partial Response (PR): >/= to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. Responders must be on same/decreasing doses of dexamethasone.
  Stable/No Response: Does not qualify for CR, PR, or progression.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over BL if no decrease), OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
  ORR = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Poly-ICLC Recurrent Gliomas: Poly-ICLC 20ug/kg 3 times a week 4 week cycles (Monday-Wednesday-Friday)
  Intramuscular injection
  Drug Poly-ICLC
  poly ICLC
Arm/Group | Poly-ICLC Recurrent Gliomas
Number analyzed (Participants) | 45
Participants | 5

2. Primary Outcome: Percentage of Participants With Progression Free Survival
Description: Participants evaluated from date of study entry to the 6 month scan for progression
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Poly-ICLC Recurrent Gliomas
Number analyzed (Participants) | 45
percentage of participants | 24

3. Secondary Outcome: Number if Participants With Grade 3 and 4 Toxicities Associated With Poly-ICLC in Recurrent Gliomas
Description: Toxicities defined by Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Poly-ICLC Recurrent Gliomas
Number analyzed (Participants) | 45
Participants
  Dyspnea | 1
  Elevated Alanin Aminotransferase | 4
  Hypoxia | 1
  Leukopenia | 2
  Muscle Weakness | 1
  Elevated Sodium | 1
  Tremors | 2

4. Secondary Outcome: Overall Survival
Description: based on date of study entry
Time Frame: 2 years
Population: Survival time was known for all 45 patients and 13 patients were censored as they were alive at last contact
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Poly-ICLC Recurrent Gliomas
Number analyzed (Participants) | 45
weeks | 43 [27.4 to 106]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Poly-ICLC Recurrent Gliomas
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 45/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly-ICLC Recurrent Gliomas (N=45)
fatigue (General disorders) | 28 (28)
injection site reaction (Skin and subcutaneous tissue disorders) | 3 (3)
Elevated Alanine Transferase (Investigations) | 13 (13)
Granulocytopenia (Investigations) | 7 (7)
Leukopenia (Investigations) | 13 (13)
Lymphocytopenia (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No